CLINICAL TRIAL: NCT07137052
Title: A Prospective Multi-center Clinical Study on Precise Guidance of Adaptive Radiotherapy for Nasopharyngeal Carcinomar by Multi-dimensional Molecular Imaging
Brief Title: Precise Guidance of Adaptive Radiotherapy for Nasopharyngeal Carcinomar
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Collaborators: Sun Yat-sen University (Other); Peking University Shenzhen Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Shandong Cancer Hospital and Institute (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shenzhen Yino Intelligence Technology Development Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Lin Qin, Prof., The First Affiliated Hospital of Xiamen University
Other Study IDs: XMYY-2025KY055
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Nasopharyngeal Carcinoma (NPC); PET / CT
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — At 1, 2, and 3 years after radiotherapy, complete blood counts, blood biochemistry tests, and Epstein-Barr virus testing (primarily measurement of Epstein-Barr virus deoxyribonucleic acid (DNA) copy number in blood) will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 68Ga-FAPI-LM3 & 68Ga-PD-L1 PET/CT Imaging Evaluation Cohort

SUMMARY:
This is an observational cohort study designed to (1) evaluate whether Gallium-68 (68Ga)-labeled fibroblast activation protein inhibitor ligand LM3 (68Ga-FAPI-LM3) positron emission tomography/computed tomography (PET/CT) improves the accuracy of nasopharyngeal carcinoma (NPC) staging, and (2) determine whether Gallium-68-labeled programmed death-ligand 1 (68Ga-PD-L1) PET/CT imaging parameters can provide early prediction of response to neoadjuvant immunotherapy. The study will assess the sensitivity and specificity of each tracer for staging and for predicting therapeutic response, analyze changes in tumor uptake parameters on 68Ga-FAPI-LM3 and 68Ga-PD-L1 PET/CT before and after treatment, and compare treatment efficacy and survival outcomes between patients with different degrees of residual PET uptake and between those who did and did not receive neoadjuvant immunotherapy. The primary question it aims to answer is:

Does 68Ga-FAPI-LM3 PET/CT improve the accuracy of NPC staging, and can 68Ga-PD-L1 PET/CT imaging parameters provide an early prediction of response to neoadjuvant immunotherapy?

Participants will be patients with biopsy-proven nasopharyngeal carcinoma who undergo 68Ga-FAPI-LM3 and/or 68Ga-PD-L1 PET/CT as part of clinical care or a research protocol. Tumor uptake metrics (e.g., maximum standardized uptake value (SUVmax), mean standardized uptake value (SUVmean), metabolic/volumetric indices) will be measured pre- and post-treatment; diagnostic performance (sensitivity, specificity) and associations between uptake changes and clinical outcomes (response rates, progression-free and overall survival) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex; age 18-70 years.
2. Histologically confirmed non-keratinizing nasopharyngeal carcinoma (World Health Organization (WHO) type II or III).
3. Clinical stage I-IVA (American Joint Committee on Cancer (AJCC)/Union for International Cancer Control (UICC) 8th edition) with no evidence of distant metastasis.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. No prior anti-tumor treatment for nasopharyngeal carcinoma, including radiotherapy, chemotherapy, immunotherapy, or biologic therapy.
6. No contraindications to radiotherapy or chemotherapy.
7. Adequate major organ function as defined below:

   7.1 Hematology: white blood cell (WBC) ≥ 4.0 × 10^9/L, absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L (no blood transfusion or blood products within 14 days and no use of granulocyte colony-stimulating factor (G-CSF) or other hematopoietic growth factors to correct counts);

   7.2 Biochemistry: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN); blood urea nitrogen (BUN) and serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min calculated by the Cockcroft-Gault formula.
8. Participant voluntarily agrees to join the study, signs informed consent, has good compliance, and is able to attend follow-up.

Exclusion Criteria:

1. Pathological type of keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
2. History of or concurrent other active (unresolved) malignant tumors, except for previously cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, or superficial bladder cancer.
3. Currently participating in another clinical trial.
4. Pregnant or breastfeeding women.
5. Uncontrolled cardiovascular disease, including ≥ Grade II myocardial ischemia or myocardial infarction, uncontrolled cardiac arrhythmias (including corrected QT (QTc) interval ≥ 470 ms); heart failure New York Heart Association (NYHA) class III-IV, or left ventricular ejection fraction (LVEF) < 50% on echocardiography; or myocardial infarction within the past year.
6. Other severe comorbidities such as uncontrolled hypertension, severe cerebrovascular disease, severe renal disease, uncontrolled diabetes mellitus, or other chronic wasting diseases.
7. History of substance or alcohol abuse, psychiatric illness, or lack of full or having limited civil capacity.
8. In the investigator's judgment, other familial or social factors that could force premature withdrawal from the study, or other conditions likely to affect participant safety or the collection of trial data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed nasopharyngeal carcinoma without distant metastasis who have not received any anti-tumor (anti-cancer) therapy.
Sampling Method: Non-Probability Sample
Enrollment: 732 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 yeas
PFS | 3 years

IPD SHARING:
Plan to Share IPD: Undecided